CLINICAL TRIAL: NCT02792491
Title: Phase II Prospective Trial of Addition of Rituximab to Reduced Dose CHOP Chemotherapy in DLBC L Patients Aged 65 Years and Over
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Ho-Jin Shin, Division of hematology-oncology, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Elderly RD_R-CHOP
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced dose R-CHOP (Experimental): Reduced dose R-CHOP is regimen including Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone.
  In this study, Rituximab 375 mg/m2, Cyclophosphamide 600 mg/m2, Doxorubicin 30 mg/m2 and Vincristine fixed dose of 1mg will be administrated through intravenous on day 1. and Prednisone 40mg will be administrated orally on day 1-5. This chemotherapy will be repeated every 21 days.
  Interventions: Drug: Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone

INTERVENTIONS:
Drug: Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone — Reduced dose of Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone
  Other Names: R-CHOP

SUMMARY:
This is Phase II prospective trial of addition of rituximab to reduced dose CHOP chemotherapy in DLBC L patients aged 65 years and over.

DETAILED DESCRIPTION:
The body surface area(BSA) on the date of every treatment cycle may be used as the same value of baseline BSA, if change of body weight is within 10% of baseline body weight. But, if there is a change of body weight more than 10% that of baseline, BSA should be recalculated. It will be repeated every 21 days. But the change of starting date of subsequent cycle and laboratory or radiologic tests may be allowed within 4 days from the scheduled date or delay due to toxicities. The RD-RCHOP treatment will be continued up to 6-8 cycles (or 3 cycles in case of stable disease(SD) or progressive disease(PD) after the first 3cycles) with duration of 21 days. Visit windows ± 4days in Treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CD20 positive DLBCL
2. Age ≥ 65 years
3. Ann Arbor stage II, III and IV
4. No prior chemotherapy or radiotherapy for DLBCL
5. Performance status (ECOG) ≤ 2
6. At least one or more bidimensionally measurable lesion(s)

   * 2 cm by conventional CT
   * 1 cm by spiral CT skin lesion (photographs should be taken) ≥ 2 cm measurable lesion by physical examination ≥ 2 cm
7. Cardiac ejection fraction ≥ 50 % as measured by MUGA or 2DECHO without clinically significant abnormalities
8. Adequate renal function: serum creatinine level < 2 mg/dL (177 μmol/L)
9. Adequate liver functions:

   Transaminase (AST/ALT) < 3 X upper normal value (or < 5 x ULN in the presence of DLBCL involvement of the liver) Bilirubin < 2 X upper normal value (or < 5 x ULN in the presence of DLBCL involvement of the liver)
10. Adequate BM functions: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL, unless abnormalities are due to bone marrow involvement by lymphoma
11. Life expectancy more than 6 months
12. A negative serum or urine pregnancy test prior to treatment must be available both for pre-menopausal women and for women who are < 1years after the onset of menopause.
13. Informed consent

Exclusion Criteria:

1. Other subtypes NHL than DLCBL
2. Patients who transformed follicular lymphoma or other indolent lymphoma
3. Primary Central Nervous System (CNS) DLBCL
4. CNS involvement by lymphoma or any evidence of spinal cord compression. Brain CT/MRI is only mandatory (within 4 weeks) in case of clinical suspicion of CNS involvement by lymphoma. Patients who have only had prophylactic intrathecal chemotherapy against CNS disease are eligible.
5. Patients with a known history of HIV seropositivity or HCV (+). Patients who have HBV (+) are eligible. However, primary prophylaxis using antiviral agents (i.e. lamivudine) is recommended for HBV carrier to prevent HBV reactivation during whole treatment period.
6. Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
7. Pregnant or lactating women, women of childbearing potential not employing adequate contraception
8. Other serious illness or medical conditions i. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry ii. History of significant neurologic or psychiatric disorders including dementia or seizures iii. Active uncontrolled infection (viral, bacterial or fungal infection) iv. Other serious medical illnesses
9. Known hypersensitivity to any of the study drugs or its ingredients (i.e., hypersensitivity to Polysorbate 20, CHO cell products, or recombinant human antibodies)
10. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
3 year progression free survival rate | Time between the date of treatment start and the date of death due to any cause or date of disease progression, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
Overall response rate | Until the disease progression (maximum 3 years after completion of treatment, assessed up to 36 months(
Overall survival | Time between the date of treatment start and the date of death due to any cause or date of disease progression, whichever came first, assessed up to 36 months
Toxicity profile | From the date of first drug administration until the date of the 30th days

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Jin Ho-Jin, Principal Investigator — Pusan National University Hospital

IPD SHARING:
Plan to Share IPD: Yes
We will share collected data with principal investigators in Korea.